CLINICAL TRIAL: NCT05318183
Title: Assessing Gut Microbiota Mediated Health Outcomes of Whole Wheat and Its Major Bioactive Components
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Richard Bruno, Principal Investigator, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2021H0347
Record Dates: First submitted 2022-03-23; First posted 2022-04-08 (Actual); Results first posted 2025-08-29 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: PreDiabetes; Dysbiosis; Endotoxemia; Inflammation
Keywords: Gut microbiota; Microbiome; Metabolomics; Prediabetes; Glycemic response; Intestinal permeability; Gut dysbiosis; Microbiome metabolism; Whole Wheat; Phytochemicals
MeSH Terms: conditions — Prediabetic State; Dysbiosis; Endotoxemia; Inflammation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive 4 servings per day of whole wheat bread (WWB) or white bread (WB) for 2 weeks. During each study arm, participants will be provided eucaloric standardized diets that are devoid of whole wheat products, probiotic-containing foods, and fermented foods. Before and after each study arm, a fasting blood sample and fecal sample will be obtained for metabolomic and clinical measures. Anthropometric measurements and blood pressure will be assessed at days 0, 7, and 14 of each study arm. On day 14, participants will complete an oral glucose tolerance test (OGTT) with collection of blood samples every 30 minutes for 3 hours and a simultaneous gut permeability test that entails ingesting non-digestible sugar probes and subsequent 24-h collection of urine. Upon completion of these procedures, participants will undergo a ~1 month washout before repeating the study identically, with the crossover to the alternate bread diet.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole Wheat Bread (Experimental): Participants consuming 128 g of whole wheat bread (4 slices of bread) daily for two weeks
  Interventions: Other: Whole Wheat Bread
- White Bread (control) (Placebo Comparator): Participants consuming 128 g of white bread (4 slices of bread) daily for two weeks
  Interventions: Other: White Bread (control)

INTERVENTIONS:
Other: Whole Wheat Bread — Standardized whole wheat bread (128 g daily)
  Arms: Whole Wheat Bread
Other: White Bread (control) — Standardized white bread (128 g daily)
  Arms: White Bread (control)

SUMMARY:
This study will investigate the gut microbiota-mediated effects of whole wheat consumption on human health in adults with pre-diabetes. Participants will complete two phases of intervention in random order in which they will consume either whole wheat bread (4 servings) or white bread a day for two weeks prior to collecting specimens (stool, urine, and plasma/serum).

DETAILED DESCRIPTION:
Accumulating clinical evidence suggests positive effects of whole grain on cardiometabolic risk. However, outcomes of controlled trials indicate that substantial interpersonal variation occurs in these studies with regard to glucose homeostasis, with some persons being unaffected and others experiencing glucose-lowering effects due to whole wheat bread consumption. Whole grain (whole wheat) contains bioactive phytochemicals in addition to its well-recognized fiber content, and these constituents have not received adequate study to inform dietary recommendations. The objective of this study is to investigate the glucose-lowering effects of whole wheat bread in persons with prediabetes using multi-omics platforms that can provide an understanding of the complex interactions among the gut microbiome, gut metabolome, host metabolome, and gut barrier function. The hypothesis is that gut microbial metabolism of whole wheat and its major bioactive components is a determining factor of human health benefits. This will be tested by conducting a randomized, controlled crossover trial in persons with pre-diabetes who follow a controlled diet containing whole wheat bread or white bread for 2-weeks. Outcomes are expected to significantly advance an understanding of personalized, gut microbiome-mediated approaches in individuals with pre-diabetes to help guide dietary recommendations of whole wheat intake. In addition, novel evidence that maps out the differential functions of diverse genus/species of microbiota to biotransform whole wheat nutrients into more bioactive metabolites are expected.

ELIGIBILITY:
Inclusion Criteria:

* Fasting blood glucose between 100-125 mg/dL
* BMI of 30-35 kg/m2

Exclusion Criteria:

* History of liver disease, cardiovascular disease, overt diabetes, or cancer
* Prescribed medications for hyperglycemia or dyslipidemia
* Use of dietary supplements, prebiotics, or probiotics
* Usage of antibiotics or anti-fungals within 3 months prior to enrollment
* Smoker
* Alcohol consumption greater than 2 drinks per day
* Aerobic exercise greater than 5 hours per week
* Pregnancy or fertility treatments
* History of chronically active inflammatory or neoplastic disease in 3 years prior to enrollment
* History of chronic gastrointestinal disorder including diarrhea, inflammatory bowel disease, celiac disease; coagulation disorders, chronic immunosuppressive medication usage
* History of myocardial infarction or cerebrovascular accident within 6 months prior to participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2026-05-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bruno, PhD, RD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Background] Cao S, Pierson JT, Bond AH, Zhang S, Gold A, Zhang H, Zamary KM, Moats P, Teegarden MD, Peterson DG, Mo X, Zhu J, Bruno RS. Intestinal-level anti-inflammatory bioactivities of whole wheat: Rationale, design, and methods of a randomized, controlled, crossover dietary trial in adults with prediabetes. Nutr Res. 2024 Nov;131:83-95. doi: 10.1016/j.nutres.2024.09.010. Epub 2024 Sep 18. PMID 39378659

RESULTS

PARTICIPANT FLOW:
Groups:
- Whole Wheat Bread, Then White Bread: Participants consuming 128 g of whole wheat bread (4 slices of bread) daily for two weeks, followed by a 2-week washout period, then consumed white bread daily for 2 weeks.
  Whole Wheat Bread: Standardized whole wheat bread (128 g daily)
- White Bread (Control), Then Whole Wheat Bread: Participants consumed 128 g of white bread (4 slices of bread) daily for two weeks, followed by a 2-week washout period, and then consumed whole wheat bread daily for an additional 2 weeks.
  White Bread (control): Standardized white bread (128 g daily)
Period: First Intervention (2 Weeks)
Arm/Group | Whole Wheat Bread, Then White Bread | White Bread (Control), Then Whole Wheat Bread
Started | 25 | 24
Completed | 21 | 21
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 2 | 0
Period: Washout (2 Weeks)
Arm/Group | Whole Wheat Bread, Then White Bread | White Bread (Control), Then Whole Wheat Bread
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0
Period: Second Intervention (2 Weeks)
Arm/Group | Whole Wheat Bread, Then White Bread | White Bread (Control), Then Whole Wheat Bread
Started | 21 | 21
Completed | 21 | 18
Not Completed | 0 | 3
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics of participants with prediabetes at screening.
Groups:
- Overall: Baseline characteristics of participants at screening
Arm/Group | Overall
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 39
BMI [Mean (Standard Deviation); unit: kg/m^2] | 34.7 (5.2)
Fasting plasma glucose [Mean (Standard Deviation); unit: mg/dL] | 108.7 (6.3)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 122.6 (10.3)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 81.9 (7.5)
Waist circumference [Mean (Standard Deviation); unit: cm] | 106.1 (12.3)

OUTCOME MEASURES:

1. Primary Outcome: Plasma Glucose
Description: Data are biomarker area under the time-concentration curve (0-3 hours) on day 14
Time Frame: Day 14 (0, 30, 60, 90, 120, 150, 180 minutes post oral glucose tolerance test)
Measure: Mean (Standard Error); unit: mg/dL x min
Arm/Group | Whole Wheat Bread | White Bread (Control)
Number analyzed (Participants) | 39 | 39
mg/dL x min | 4092.15 (597.81) | 5622.96 (644.59)

2. Secondary Outcome: Plasma Insulin
Description: Data are biomarker fasting concentrations
Time Frame: Day 14
Measure: Mean (Standard Error); unit: uIU/mL
Arm/Group | Whole Wheat Bread | White Bread (Control)
Number analyzed (Participants) | 39 | 39
uIU/mL | 18.9 (2.8) | 16.0 (1.6)

3. Secondary Outcome: Plasma Glucose
Description: Data are biomarker fasting concentrations.
Time Frame: Day 14
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Whole Wheat Bread | White Bread (Control)
Number analyzed (Participants) | 39 | 39
mg/dL | 93.5 (2.6) | 85.6 (2.3)

4. Secondary Outcome: Serum C-reactive Protein
Description: Data are the biomarker serum concentration of C-reactive protein.
Time Frame: Day 14
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Whole Wheat Bread | White Bread (Control)
Number analyzed (Participants) | 39 | 39
mg/dL | 0.47 (0.1) | 0.53 (0.1)

5. Secondary Outcome: Serum Tumor Necrosis Factor Alpha
Description: Data are biomarker serum tumor necrosis factor alpha concentrations.
Time Frame: Day 14
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Whole Wheat Bread | White Bread (Control)
Number analyzed (Participants) | 39 | 39
pg/mL | 6.39 (1.0) | 5.63 (0.6)

6. Secondary Outcome: Serum Interleukin-6
Description: Data are biomarker serum interleukin-6 concentrations.
Time Frame: Day 14
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Whole Wheat Bread | White Bread (Control)
Number analyzed (Participants) | 39 | 39
pg/mL | 1.88 (0.2) | 1.94 (0.2)

7. Secondary Outcome: Fecal Calprotectin
Description: Data are biomarker fecal concentrations.
Time Frame: Day 14
Measure: Mean (Standard Error); unit: ug/g
Arm/Group | Whole Wheat Bread | White Bread (Control)
Number analyzed (Participants) | 39 | 39
ug/g | 32.8 (4.6) | 35.84 (5.2)

8. Secondary Outcome: Fecal Myeloperoxidase
Description: Data are biomarker fecal concentrations.
Time Frame: Day 14
Measure: Mean (Standard Error); unit: ng/g
Arm/Group | Whole Wheat Bread | White Bread (Control)
Number analyzed (Participants) | 39 | 39
ng/g | 116 (31.5) | 157 (20.9)

9. Secondary Outcome: Urine Lactulose/Mannitol
Description: Data are the 24-hour urinary excretion ratio of lactulose relative to mannitol collected 0-5 h following the digestion of non-digestible sugar probes.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

10. Secondary Outcome: Urine Sucralose/Erythritol
Description: Data are the sucralose/erythritol ratio measured in urine collected 6-24 h following the digestion of non-digestible sugar probes.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

11. Secondary Outcome: Serum Endotoxin
Description: Data are biomarker fasting concentrations.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

12. Secondary Outcome: Serum Myeloperoxidase
Description: Data are biomarker serum concentrations.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

13. Secondary Outcome: Level of Toll-like Receptor 4 Gene Expression
Description: Data are expression of toll-like receptor 4 gene from peripheral blood mononuclear cells.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

14. Secondary Outcome: Myeloid Differentiation Factor 88 Gene Expression
Description: Expression of myeloid differentiation factor 88 gene from peripheral blood mononuclear cells.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

15. Secondary Outcome: Tumor Necrosis Factor Alpha Gene Expression
Description: Expression of tumor necrosis factor alpha gene from peripheral blood mononuclear cells.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

16. Secondary Outcome: p65 Subunit of Nuclear Factor Kappa B Gene Expression
Description: Expression of p65 subunit of nuclear factor kappa B gene from peripheral blood mononuclear cells.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

17. Secondary Outcome: Interleukin-6 Gene Expression
Description: Expression of interleukin-6 gene from peripheral blood mononuclear cells.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

18. Secondary Outcome: Interleukin-8 Gene Expression
Description: Expression of interleukin-8 gene from peripheral blood mononuclear cells.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

19. Secondary Outcome: Myeloperoxidase Gene Expression
Description: Expression of myeloperoxidase gene from peripheral blood mononuclear cells.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

20. Secondary Outcome: Monocyte Chemoattractant Protein-1 Gene Expression
Description: Expression of monocyte chemoattractant protein-1 gene from peripheral blood mononuclear cells.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

21. Secondary Outcome: Fecal Butyrate
Description: Data are biomarker fecal concentrations.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

22. Secondary Outcome: Fecal Acetate
Description: Data are biomarker fecal concentrations.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

23. Secondary Outcome: Fecal Propionate
Description: Data are biomarker fecal concentrations.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

24. Secondary Outcome: Fecal Isobutyric Acid
Description: Data are biomarker fecal concentrations.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

25. Secondary Outcome: Fecal Isovaleric Acid
Description: Data are biomarker fecal concentrations of isovaleric acid.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

26. Secondary Outcome: Serum Alkylersorcinols
Description: Data are biomarker serum concentrations of alkylresorcinol and alkylresorcinol derivatives.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

27. Secondary Outcome: Serum Benoxazinods
Description: Data are biomarker serum concentrations of benoxazinoids and benoxazinoids derivatives.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

28. Secondary Outcome: Serum Phenolic Compounds
Description: Data are biomarker serum concentrations of phenolic compounds and phenolic derivatives.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

29. Secondary Outcome: Fecal Alkylresorcinols
Description: Data are biomarker fecal concentrations of alkylresorcinols and alkylresorcinol derivatives.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

30. Secondary Outcome: Fecal Benoxazinoids
Description: Data are biomarker fecal concentrations of benoxazinoids and benoxazinoids derivatives.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

31. Secondary Outcome: Fecal Phenolic Compounds
Description: Data are fecal concentrations of phenolic compounds and phenolic derivatives.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

32. Other Pre Specified Outcome: Plasma Triglyceride
Description: Data are biomarker fasting plasma concentrations.
Time Frame: Day 0, Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

33. Other Pre Specified Outcome: Plasma Cholesterol Levels
Description: Data are biomarker fasting plasma concentrations.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

34. Other Pre Specified Outcome: Plasma HDL-cholesterol
Description: Data are biomarker fasting plasma concentrations.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

35. Other Pre Specified Outcome: Serum Alanine Transaminase
Description: Data are biomarker serum concentrations of alanine transaminase.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

36. Other Pre Specified Outcome: Serum Interleukin-8
Description: Data are biomarker serum interleukin-8 concentrations.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

37. Other Pre Specified Outcome: Gut Microbiota Alpha-diversity Indices
Description: Alpha-diversity will be determined based on the Shannon-Wiener diversity index. Fecal microbiota assessments and the subsequent determinations of alpha-diversity.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

38. Other Pre Specified Outcome: Gut Microbiota Beta-diversity Indices
Description: Beta-diversity will be determined based on the Bray-Curtis diversity index. Fecal microbiota assessments and the subsequent determinations of beta-diversity.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

39. Other Pre Specified Outcome: Gut Microbiota Relative Abundance
Description: Gut microbiota relative abundance (percent order, genus, and species level) will be measured in fecal samples.
Time Frame: Day 14
Reporting Status: Not Posted, anticipated posting 2026-05

ADVERSE EVENTS:
Time Frame: 3-months
Arm/Group | Whole Wheat Bread | White Bread (Control)
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/45
Other Adverse Events (participants affected / at risk) | 0/46 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT05318183/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/83/NCT05318183/ICF_001.pdf